CLINICAL TRIAL: NCT04167059
Title: Implementing Telehealth Support to Increase Physical Activity in Girls and Women With Rett Syndrome
Brief Title: Telehealth Support to Increase Physical Activity in Rett Syndrome
Acronym: ActivRett
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Telethon Kids Institute (Other)
Collaborators: Rigshospitalet, Denmark (Other); Ariel University (Other); University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGS0000003371
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Rett Syndrome
Keywords: Sedentary behaviour; Physical activity; Quality of life; Telehealth
MeSH Terms: conditions — Rett Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: We are using a waitlist controlled trial study design. Group membership will be determined using a concealed allocation randomisation after the baseline assessment. The 'immediate treatment' group will receive the 12-week intervention period following the assessment at baseline followed by a 12 week non-intervention period. The 'waitlist control' group receive no intervention in the first 12 week period and will then receive the intervention in the second 12 week period.
Masking Description: We note that our primary outcomes of sedentary behaviours and physical activity will be measured objectively by physical activity devices.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist-Control Group (Experimental): The 'waitlist control' group will receive the 12-week non-intervention period first, followed by 12 week intervention period.
  Interventions: Behavioral: Telehealth-delivered participation strategies to increase physical activity
- Immediate Treatment (Experimental): The 'immediate treatment' group will receive the 12-week intervention period first, followed by 12 week non-intervention period.
  Interventions: Behavioral: Telehealth-delivered participation strategies to increase physical activity

INTERVENTIONS:
Behavioral: Telehealth-delivered participation strategies to increase physical activity — Therapists and primary caregivers will meet online on 6 occasions at fortnightly intervals over a 12 week period. Sessions will enable the development of strategies that will aim to increase the amount the participant stands and walks. Throughout, the therapists and primary caregivers will discuss physical activity needs, determine relevant activities, modify the program as necessary and plan additional goals.

SUMMARY:
This study will recruit families with a daughter with Rett syndrome living in either Australia, Denmark or Israel, and thereafter deliver individually designed participation programs using telehealth strategies. We will evaluate the effectiveness of the programs on reducing sedentary behaviours, increasing physical activity and increasing quality of life.

DETAILED DESCRIPTION:
This project will implement two intertwined strategies that will build the capacity of the carer, clinical and therapy communities to support physical activity in Rett syndrome. Individuals with Rett syndrome experience difficulties with movement and this can make it difficult to participate in regular physical activity. Individuals with Rett syndrome need support to participate in physical activities and it is important to work with primary caregivers when developing strategies to support physical activity. We will conduct a clinical trial that tests the effectiveness of working with primary caregivers to develop strategies suitable to their lives that aim to increase participation in physical activity in the individual with Rett syndrome whom they support. We will use a clinical trial design and work with primary caregivers using Telehealth. We will test whether this approach decreases sedentary time and increases physical activity. We will also test if there are changes in the sleep, behaviour and quality of life. We aim to recruit 60 families for this study, 26 of whom will live in Australia. Data from the three sites will be pooled for a stronger analysis. We acknowledge that physical activity can be associated with a fall and therefore our program will be developed with the primary caregiver to be suitable for their lives and capacity to provide support. However, by practicing more activity, the individuals with Rett syndrome could be stronger and risks of falling could be reduced. The risks for the individual with Rett syndrome are therefore low. To let the Rett syndrome community know our results, we will then develop an online resource documenting the physical activity program and the evidence available to support it, and this will be freely available to families, carers and therapists wherever they live in the world.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed Rett syndrome
* Able to stand (with or without assistance)
* Live in Australia, Denmark or Israel

Exclusion Criteria:

* Individuals who have had spinal fusion over the previous 12 months
* Individuals who have had lower extremity orthopaedic surgery over the previous 6 months

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Average daily uptime (%) | Average over 4 days, data capture at baseline, after 12 weeks and after 24 weeks
  Percentage of time spent active (uptime) over total awake time, measured with an ActivPAL
Average daily step count | Average over 4 days, data capture at baseline, after 12 weeks and after 24 weeks
  Number of daily steps measured by Stepwatch Activity Monitor

SECONDARY OUTCOMES:
Sleep quality | Parent caregiver recall over previous month, data capture at baseline, after 12 weeks and after 24 weeks
  Sleep Disturbance Scale for Children.
Behaviour | Parent caregiver recall over previous month, data capture at baseline, after 12 weeks and after 24 weeks
  Rett Syndrome Behaviour Scale
Child Quality of Life | Parent caregiver recall over previous month, data capture at baseline, after 12 weeks and after 24 weeks
  Quality of Life Inventory-Disability (QI-Disability)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Downs, PhD, Principal Investigator — Telethon Kids Institute
Locations (2):
- Center for Rett Syndrom, Rigshospitalet, Copenhagen, Denmark
- Ari'el University, Ari’el, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Downs J, Lotan M, Elefant C, Leonard H, Wong K, Buckley N, Stahlhut M. Implementing telehealth support to increase physical activity in girls and women with Rett syndrome-ActivRett: protocol for a waitlist randomised controlled trial. BMJ Open. 2020 Dec 29;10(12):e042446. doi: 10.1136/bmjopen-2020-042446. PMID 33376177